CLINICAL TRIAL: NCT05896865
Title: Radiotherapy Dose Adaptation Based on Tumor Biology in Patients With cN2b-N3 Breast Cancer: Non-randomized Phase II, Prospective Single Arm Study Clinical Trial
Brief Title: Radiotherapy Dose Adaptation Based on Tumor Biology in Patients With cN2b-N3 Breast Cancer
Acronym: RADAPT-N3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Haeyoung Kim, Associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01-012
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative radiation therapy to breast / chest wall and regional lymph node area (Experimental): Patient achieved complete response after neoadjuvant chemotherapy will receive postoperative radiation therapy with dose of 42.4 Gy in 16 fractions to whole breast / chest wall and regional lymph node area. Internal mammary or supraclavicular lymph node area boost will be simultaneously delivered with total dose of 53.6 Gy in 16 fractions.
  Patient with partial response, stable disease, or progressive disease after neoadjuvant chemotherapy will receive postoperative radiation therapy with dose of 42.4 Gy in 16 fractions to whole breast / chest wall and regional lymph node area. Internal mammary or supraclavicular lymph node area boost will be simultaneously delivered with total dose of 56.0 Gy in 16 fractions.
  Interventions: Radiation: Whole breast / chest wall & regional lymph node irradiation; Radiation: Internal mammary or supraclavicular lymph node boost

INTERVENTIONS:
Radiation: Whole breast / chest wall & regional lymph node irradiation — Whole breast / chest wall and corresponding regional lymph node irradiation with dose of 42.4 Gy in 16 fractions
Radiation: Internal mammary or supraclavicular lymph node boost — Simultaneous boost to Internal mammary or supraclavicular lymph node area with dose of total 53.6 Gy or 56.0 Gy in 16 fractions, depending on the response after neoadjuvant chemotherapy

SUMMARY:
The purpose of the study is to evaluate treatment outcomes of breast cancer with internal mammary or supraclavicular lymph node metastasis according to total radiation dose of postoperative radiation therapy differentiated by tumor response to neoadjuvant chemotherapy.

The main questions it aims to answer are:

* 5-year disease-free survival
* 5-year overall survival
* 5-year locoregional recurrence
* Adverse events after radiation therapy
* Quality of life

Participants will be assessed by multi-dimensional methods before and after radiotherapy:

* Disease status evaluation including physical and radiological examination
* Quality of life assessment with questionnaires (BREAST-Q)
* Adverse event assessment according to CTCAE version 5.0

ELIGIBILITY:
Inclusion Criteria:

* Female with age 19 or older
* Metastasis to internal mammary and/or supraclavicular lymph nodes, assessed by radiological exams and/or biopsy
* Underwent neoadjuvant chemotherapy
* Pathologic confirmation of invasive breast cancer treated with breast conserving surgery or mastectomy
* Eastern Cooperative Oncology Group performance status 0-2
* Informed consent

Exclusion Criteria:

* Previous history of radiation therapy to the chest
* Distant metastasis

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2028-03-16 (Estimated); Study Completion 2030-03-16 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival | 5 years from the initiation of the radiation therapy
  The event for disease-free survival is defined as any disease recurrence or breast cancer-related death

SECONDARY OUTCOMES:
5-year overall survival | 5 years from the initiation of the radiation therapy
  The event for overall survival is defined as death of patient with any cause.
5-year locoregional recurrence | 5 years from the initiation of the radiation therapy
  The event for locoregional recurrence is defined as disease recurrence in irradiated breast / chest wall and/or regional lymph node area including internal mammary and supraclavicular lymph node area.
Adverse events | 5 years from the initiation of the radiation therapy
  Adverse events after radiation therapy is graded according to CTCAE version 5.0.
Quality of life (BREAST-Q™) | 5 years from the initiation of the radiation therapy
  Quality of life is assessed by BREAST-Q™ questionnaires. Each score from BREAST-Q™ scales ranges from 0 to 100. Higher scores reflect a better outcome except Cancer Worry scale.

CONTACTS AND LOCATIONS:
Overall Officials: Haeyoung Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No